CLINICAL TRIAL: NCT02167204
Title: Cellular Proliferation Imaging Using [18F] Fluorothymidine (FLT) Positron Emission Tomography (PET) in Brain Tumors
Brief Title: 18F-FLT PET/CT in Measuring Cell Proliferation in Patients With Brain Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 7754; NCI-2013-02162 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 7754 (Other: Fred Hutch/University of Washington Cancer Consortium); P01CA042045 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Metastatic Malignant Neoplasm in the Brain; Primary Brain Neoplasm; Recurrent Brain Neoplasm
MeSH Terms: conditions — Brain Neoplasms | interventions — alovudine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnostic (18F-FLT PET/CT) (Experimental): Patients undergo 18F-FLT PET/CT at baseline (pre-therapy), mid-therapy, completion of therapy, and 1 year after completion of therapy or time of suspected recurrence.
  Interventions: Procedure: Computed Tomography; Radiation: Fluorothymidine F-18; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo 18F-FLT PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT SCAN; tomography
Radiation: Fluorothymidine F-18 — Undergo 18F-FLT PET/CT
  Other Names: 18F-FLT; 3'-Deoxy-3'-(18F) Fluorothymidine; 3'-deoxy-3'-[18F]fluorothymidine; Fluorothymidine F 18
Procedure: Positron Emission Tomography — Undergo 18F-FLT PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This pilot clinical trial studies fluorine F 18 fluorothymidine (FLT) positron emission tomography (PET)/computed tomography (CT) in measuring cell proliferation in patients with brain tumors. Comparing results of diagnostic procedures done before, during, and after treatment may help doctors measure tumor growth and plan the best treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Using FLT PET/CT as a measure of cellular proliferation, assess tissue proliferation in disease sites of brain tumor patients before therapy (surgery, chemotherapy or radiotherapy or any combination of these).

II. Determine level of change in cellular proliferation compared with baseline (scan 1) in brain tumors at mid-therapy (scan 2), after completion of therapy (scan 3) and in the clinical follow-up period (scan 4), when possible.

III. Correlate levels of cellular proliferation measured by FLT PET/CT at baseline and treatment-induced changes in brain tumor proliferation with clinical response status (clinical categories are complete remission, lesser degrees of response/stable disease, and no response).

SECONDARY OBJECTIVES:

I. Assess spatial heterogeneity of FLT uptake to identify local differences in brain tumor disease burden.

OUTLINE:

Patients undergo 18F-FLT PET/CT at baseline (pre-therapy), mid-therapy, completion of therapy, and 1 year after completion of therapy or time of suspected recurrence.

After completion of study, patients are followed for up to 7 years.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis or suspected diagnoses of brain tumor (primary, recurrent, or metastatic) by standard clinical diagnosis such as pathology or imaging
* Planned for treatment with radiation, chemotherapy and surgical resection or any of these treatment strategies combined

Exclusion Criteria:

* Inability to provide informed consent
* Pregnancy
* Inability to lie still for the imaging study
* Weight over 350 lbs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-11; Primary Completion 2019-01-21 (Actual); Study Completion 2019-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Rockhill, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic (18F-FLT PET/CT)
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (18F-FLT PET/CT)
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 53.5 [34.8 to 69.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Measure of FLT Flux
Description: The percentage change in the kinetic model parameter of FLT flux (Ki) was recorded. Ki is estimated from parameters derived by fitting the FLT input function and the total blood activity curve to the tissue time-activity curve data.
Time Frame: Baseline to up to 1 year after completion of treatment
Population: 4 patients had 2 scans, 2 patients had 3 scans
Measure: Median (Full Range); unit: percent change
Groups:
- 2 Diagnostic (18F-FLT PET/CT)Scans: Patients completing two 18F-FLT PET/CT scans - at baseline (pre-therapy) and mid-therapy
- 2 or 3 Diagnostic (18F-FLT PET/CT) Scans: Patients completing two or three 18F-FLT PET/CT scans - at baseline (pre-therapy) and mid-therapy and completion of therapy
Arm/Group | 2 Diagnostic (18F-FLT PET/CT)Scans | 2 or 3 Diagnostic (18F-FLT PET/CT) Scans
Number analyzed (Participants) | 6 | 6
percent change | -4 [-48 to 33] | 3 [-48 to 100]

2. Primary Outcome: Percentage Change in Measure of Reflecting Transport
Description: The percentage change in the kinetic model parameter of FLT transport (K1) was recorded. K1 is defined as the transfer of FLT from blood into tissue (tumor).
Time Frame: Baseline to up to 1 year after completion of treatment
Population: 4 patients had 2 scans and 2 had 3 scans.
Measure: Median (Full Range); unit: percent change
Groups:
- 2 Diagnostic (18F-FLT PET/CT) Scans: Patients completing two 18F-FLT PET/CT scans - at baseline (pre-therapy) and mid-therapy
- 2 or 3 Diagnostic (18F-FLT PET/CT) Scans: Patients completing three 18F-FLT PET/CT scans - at baseline (pre-therapy) and mid-therapy and completion of therapy
Arm/Group | 2 Diagnostic (18F-FLT PET/CT) Scans | 2 or 3 Diagnostic (18F-FLT PET/CT) Scans
Number analyzed (Participants) | 6 | 6
percent change | -11 [-44 to 130] | -11 [-44 to 130]

3. Primary Outcome: Percentage Change in Measure of Standard Uptake Value
Description: The percentage change in the maximum standard uptake value (SUVmax) was recorded. SUVmax is defined as the amount of FLT uptake in a lesion.
Time Frame: Baseline to up to 1 year after completion of treatment
Population: 4 patients had 2 scans, 2 patients had 3 scans
Measure: Median (Full Range); unit: percent change
Groups:
- 2 Diagnostic (18F-FLT PET/CT) Scans: Patients undergo two 18F-FLT PET/CT at baseline (pre-therapy) and mid-therapy
- 2 or 3 Diagnostic (18F-FLT PET/CT) Scans: Patients undergo three 18F-FLT PET/CT at baseline (pre-therapy), mid-therapy and completion of therapy
Arm/Group | 2 Diagnostic (18F-FLT PET/CT) Scans | 2 or 3 Diagnostic (18F-FLT PET/CT) Scans
Number analyzed (Participants) | 6 | 6
percent change | -14 [-74 to 20] | -10 [-74 to 104]

4. Primary Outcome: Survival
Description: Time from study entry to death will be recorded
Time Frame: Up to 7 years
Population: All patients with at least one 18F-FLT/CT study
Measure: Median (Full Range); unit: months
Arm/Group | Diagnostic (18F-FLT PET/CT)
Number analyzed (Participants) | 9
months | 23.2 [5.4 to 200.4]

5. Primary Outcome: Clinical Response Assessed Using Revised Assessment in Neuro-Oncology Criteria
Description: This is clinical response as assessed at physician discretion using standard of care criteria.
Time Frame: Up to 7 years
Population: Data not collected for this Outcome Measure
Arm/Group | Diagnostic (18F-FLT PET/CT)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 24 hours after injection of 18F-FLT
Description: This is an imaging study. No adverse events are expected or have been reported due to tracer injection or imaging during the 24 hour monitoring period. All deaths were due to the natural course of cancer after the time period that adverse events were collected for this study.
Arm/Group | Diagnostic (18F-FLT PET/CT)
All-Cause Mortality (participants affected / at risk) | 7/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-26): https://cdn.clinicaltrials.gov/large-docs/04/NCT02167204/Prot_SAP_000.pdf